CLINICAL TRIAL: NCT00589641
Title: Relapse Prevention for Suicidal Dually Diagnosed Youths
Acronym: CBT-RP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: UConn Health (Other); University of North Carolina, Chapel Hill (Other); University of North Carolina, Greensboro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00006806; R34MH067904 (NIH); 303-7105
Record Dates: First submitted 2007-12-31; First posted 2008-01-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2010-06

CONDITIONS: Suicide, Attempted; Suicide, Ideation; Depression; Substance Abuse
Keywords: adolescents; suicidal ideation and behavior; depression; substance abuse
MeSH Terms: conditions — Suicide, Attempted; Suicide; Depression; Substance-Related Disorders; Suicidal Ideation; Behavior | interventions — Secondary Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT-RP + Enhanced TAU (Experimental): CBT-RP augmenting relapse prevention intervention, in addition to enhanced treatment as usual, monthly check-ins, and monitoring
  Interventions: Behavioral: CBT-RP (relapse prevention) + Enhanced TAU
- Enhanced TAU (Treatment as Usual) (Active Comparator): Treatment as usual in the community, monthly monitoring regarding service use and needs, monitoring
  Interventions: Behavioral: Enhanced TAU Alone

INTERVENTIONS:
Behavioral: CBT-RP (relapse prevention) + Enhanced TAU — CBT-RP is an 20-week augmenting intervention. CBT-RP is based primarily on Alan Marlatt's cognitive behavioral relapse prevention model for substance abuse, but also includes motivational interviewing and mindfulness meditation approaches. Sessions are twice a week in first week, then weekly thereafter, with tapering to biweekly in the last 8 weeks depending on improvement. Participants also receive treatment as usual, and monthly check-ins regarding treatment use.
  Arms: CBT-RP + Enhanced TAU
Behavioral: Enhanced TAU Alone — Treatment as usual in the community, monthly check-ins regarding treatment use or needs, and monitoring
  Arms: Enhanced TAU (Treatment as Usual)

SUMMARY:
The purpose of this study is to develop, refine, and pilot test an augmenting cognitive behavior relapse prevention intervention (CBT-RP) for suicidal, depressed, and alcohol/substance abusing adolescents. No hypotheses are being tested, but it is expected that CBT-RP in addition to treatment as usual will result in improved outcomes relative to treatment as usual alone.

DETAILED DESCRIPTION:
Suicide attempts are not only associated with increased likelihood of eventual death by suicide (Lonnqvist & Ostano, 1991), increased risk of repeat suicidal behavior (Goldston et al., 1999; Leon et al., 1989), and risk of physical injury, but suicidality is also one of the primary reasons for psychiatric emergencies and psychiatric hospitalizations (Peterson et al., 1996). Suicide attempters, particularly repeat attempters, often have histories of both depression and substance abuse problems. Cognitive behavioral interventions have been shown to have promise in the treatment of depression (Brent et al., 1997), suicidality (Henriques, Beck, & Brown, 2002), and substance use disorders in youths (Dennis et al., in press; Kaminer et al., 2002). Relapse prevention approaches have been shown to have utility with substance abusing adults (Witkiewitz & Marlatt, 2004), and conceptually are well suited for the prevention of both suicidal behavior and substance use among young people. The purpose of the research outlined in this application is therefore to develop, refine, and test a cognitive behavioral relapse prevention intervention (CBT-RP) for dually diagnosed suicidal adolescents and young adults.

The specific aims of this research are as follows:

1. To develop and refine a cognitive behavioral relapse prevention treatment manual for suicidal adolescents and young adults with comorbid depressive and substance use disorders.
2. To develop and pilot test procedures for training therapists to conduct CBT-RP. Methods for assessing therapist competence and adherence to the protocols, and certification standards will be developed and refined.
3. To assess the feasibility of CBT-RP via monitoring of rates of recruitment and retention of subjects, monitoring of therapist adherence and deviation from the protocols, and monitoring of adverse events.
4. To assess the feasibility of the assessment methods and outcome measures to be used in this study as reflected in burden in completing assessments over the course of treatment.
5. To estimate the degree of change and variability of response to CBT-RP relative to no CBT-RP as an add-on treatment to Treatment as Usual (TAU) in the community on the primary outcomes of suicidal ideation, depressive symptoms, and substance use problem severity.
6. To assess the acceptability of CBT-RP relative to no CBT-RP as an add-on treatment to TAU in the community as assessed qualitatively via exit interviews and quantitatively via ratings of patient satisfaction

There are four phases to this treatment development study: (1) initial manual and protocol development (not requiring human subject involvement); (2) piloting (and revision) of the manual by the investigators; (3) training and supervision of new therapists using the new intervention; and, (4) the pilot randomized controlled trial. We have completed the first phase of this study. Currently, we are involved in completing pilot testing and initiating training of new therapists with the protocol (n=12). A subsequent pilot randomized controlled trial will be used to examine feasibility and preliminary evidence of effects (and variability of effects) of CBT-RP as an augmenting intervention (n=36).

ELIGIBILITY:
Inclusion Criteria:

* Teenagers 13-19 living with parents, or foster parents, at least one of whom is English speaking and willing to participate
* Participation in ongoing treatment in the community (or willing to accept a referral for treatment as usually delivered in the community)
* Marijuana or alcohol use or dependence disorder
* Depressive disorder (major depression, dysthymia, depressive disorder NOS)
* High suicide risk as reflected in: (a) recent suicidal behaviors (suicide attempts, aborted attempts, interrupted attempts, or suicide plans) in last 4 weeks OR (b)lifetime history of suicidal behaviors together with current clinically significant suicidal ideation (measured on a self-report questionnaire)

Exclusion Criteria:

* Substance Dependence Disorder other than alcohol or cannabis or nicotine
* SUD severity such that higher (more intensive) level of treatment (e.g., residential, hospitalization) is needed
* Psychiatric difficulty other than substance abuse, suicidality, or depression that needs to be the primary focus of treatment (e.g., severe eating disorder or psychosis)
* Evidence of mental retardation or poor receptive vocabulary as assessed with Peabody Picture Vocabulary Test

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2005-07; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
suicide ideation and behavior | pre-treatment, 10 weeks, end of treatment, 3-month follow-up

SECONDARY OUTCOMES:
depression severity, alcohol/cannabis abuse impairment | pre-treatment, 10 weeks, end of treatment, 3 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: David B Goldston, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke Child and Family Study Center, Durham, North Carolina, United States